CLINICAL TRIAL: NCT05479773
Title: Safety and Usability of the LUMENA Non-invasive Ventilation Mask
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Inspir Labs Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 0818-21-TLV
Record Dates: First submitted 2022-07-10; First posted 2022-07-29 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Other): Treatment order:
  1) Standard NIV mask ; 2) Lumena mask without suction ; 3) Lumena mask with suction.
  Interventions: Device: Standard NIV mask; Device: Lumena NIV mask
- Group B (Other): Treatment order:
  1) Standard NIV mask ; 2) Lumena mask with suction ; 3) Lumena mask without suction.
  Interventions: Device: Standard NIV mask; Device: Lumena NIV mask
- Group C (Other): Treatment order:
  1) Lumena mask without suction ; 2) Lumena mask with suction ; 3) Standard NIV mask.
  Interventions: Device: Standard NIV mask; Device: Lumena NIV mask
- Group D (Other): Treatment order:
  1) Lumena mask with suction ; 2) Lumena mask without suction ; 3) Standard NIV mask.
  Interventions: Device: Standard NIV mask; Device: Lumena NIV mask

INTERVENTIONS:
Device: Standard NIV mask — The hospital standered NIV mask
Device: Lumena NIV mask — aerosol-reducing mask

SUMMARY:
Evaluation of the safety and efficacy of using the Lumena mask, compared to commercially-available, commonly used Oro-nasal masks.

DETAILED DESCRIPTION:
20 participants will be included in the study. The number of patients for each group is 5.

The trial is, a crossover trial, as all participants go through every one of the trial conditions, albeit in a different order, and thus every trial condition will have results of 20 patients in it eventually.

Prior to patient treatment, the subject will be informed about the study and potential risks, and will be givin written informed consent.

Prior to every inhalation and particle sampling, a baseline sample will be taken to filter possible carryovers from previous sampling.

Demographics including age, sex, DOB, height, weight and body mass index. Past medical history including smoking status, co-morbid conditions and medication use.

Vital signs before, during and after non-invasive ventilation: heart rate, respiratory rate, Tidal volume, oxygen saturation, Mode of ventilation, peak inspiratory pressure, pressure support, Ventilator type and model, Trigger sensitivity, Fio 2%, PEEP, blood pressure (invasive and/or non-invasive) and temperature.

Electrocardiogram (ECG) diagrams before and after use. Arterial blood\ Venous blood gas analysis for O2, CO2, pH and HCO3 as well as serum Lactate levels before, during and after non-invasive ventilation. A maximum of 20 ml of blood will be collected from each patient.

Room aerosol particle concertation in sizes 0.3, 0.5, 1.0 and 2.5µ. Symptoms and signs during use of non-invasive ventilation (e.g. diaphoresis, anxiety).

Estimation of patient preference of the mask - the question shall be phrased thusly: In a Which mask do you prefer? Estimation of staff comfort (an analog 1-5 scale as well as recording of verbal comments). - the question shall be phrased thusly: In a scale of 1-5, 1 being very uncomfortable to use and 5 being very comfortable, to use how would you rate the mask? Estimation of staff use - the question shall be phrased thusly: Which mask do you prefer? Estimation of patient comfort - the question will be directed to the staff member. (an analog 1-5 scale as well as recording of verbal comments) - the question shall be phrased thusly: In a scale of 1-5, 1 being very uncomfortable to use and 5 being very comfortable to use, how would you rate the patient's feeling with the experimental mask? Device related AE's will be reported by number, type, seriousness, severity and duration. All device and treatment related AEs will be captured, regardless of severity.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female adults, aged 18 years and over.
2. Suffering from hypoxemic and/or hypercarbic respiratory failure requiring non-invasive ventilation and selected by medical staff to use CPAP or BiPAP.
3. Fully concious (Glasgow Coma Scale 14-15) and able to cooperate with non-invasive ventilation.
4. Able to provide informed consent to participate in the study.
5. Have an active arterial line in place for arterial blood sampling (arterial lines will not be placed for the sole purpose of the study). Alternatively, IV line can be used.

Exclusion Criteria:

1. Age < 18 years.
2. Pregnancy.
3. Respiratory failure due to non-pulmonary pathology.
4. Presence of a contraindication to the use of non-invasive ventilation or an absolute indication for invasive ventilation.
5. Presence of a facial deformity, heavy beard or moustache which prevents a good seal between the mask and the face.
6. Hemodynamic instablity.
7. Severe upper gastrointestinal bleeding.
8. Chest trauma.
9. Claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-06-23 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-06-22 (Estimated)

PRIMARY OUTCOMES:
SPO2 | During the 30 minutes before starting the ventilation
  Precentage of SPO2 before ventilation
SPO2 | Every 20 minutes during ventilation
  Precentage of SPO2 during ventilation
SPO2 | Up to 30 minutes post ventilation
  Precentage of SPO2 post ventilation
pO2 | During the 30 minutes before starting the ventilation
  mmHg of PO2 before ventilation
pO2 | Every 20 minutes during ventilation
  mmHg of PO2 during ventilation and post ventilation
pO2 | Up to 30 minutes post ventilation
  mmHg of PO2 post ventilation
pCO2 | During the 30 minutes before starting the ventilation
  pCO2 before ventilation measured in mmHg
pCO2 | Every 20 minutes during ventilation
  pCO2 during ventilation measured in mmHg
pCO2 | Up to 30 minutes post ventilation
  pCO2 post ventilation measured in mmHg
pH | During the 30 minutes before starting the ventilation
  logarithmic units of pH before ventilation
pH | Every 20 minutes during ventilation
  logarithmic units of pH during ventilation
pH | Up to 30 minutes post ventilation
  logarithmic units of pH post ventilation
HCO3 | During the 30 minutes before starting the ventilation
  HCO3 before ventilation measured in mEq/L
HCO3 | Every 20 minutes during ventilation
  HCO3 during ventilation measured in mEq/L
HCO3 | Up to 30 minutes post ventilation
  HCO3 post ventilation measured in mEq/L
Serum Lactate | During the 30 minutes before starting the ventilation
  Serum Lactate before ventilation measured in mmol/Lit
Serum Lactate | Every 20 minutes during ventilation
  Serum Lactate during ventilation measured in mmol/Lit
Serum Lactate | Up to 30 minutes post ventilation
  Serum Lactate post ventilation measured in mmol/Lit
Respiratory Rate | during ventilation
  Measuring of Respiratory Rate in breaths per minute, during ventilation
Adverse Events | From date of study randomization until the end of treatment per each patient, up to 30 min post ventilation
  Number of patients related Adverse Events as assessed by CTCAE v5.0

SECONDARY OUTCOMES:
Room aerosol concentration | Before ventilation and during ventilation
  Room aerosol concentration during usage of the Lumena for particle 0.3, 0.5, 1.0 and 2.5 Microns in units of parts per cubic meter of air
Use comfort | Up up 1 hour post ventilation
  Patient assesment of use comfort of the worn mask, in units of 1 to 5 with 5 being the highest.
Use comfort | Up up 1 hour post ventilation
  Staff member assesment of use comfort of the worn mask, in units of 1 to 5 with 5 being the highest.

CONTACTS AND LOCATIONS:
Overall Officials: Nimrod Adi, Mr, Principal Investigator — Head of ICU
Locations (1):
- Tel Aviv Sourasky Medical Center, Ichilov, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-01-01): https://cdn.clinicaltrials.gov/large-docs/73/NCT05479773/Prot_002.pdf